CLINICAL TRIAL: NCT07106359
Title: A Randomized Controlled Pilot Trial of a Behavioral Intervention to Increase Uptake of Genetic Services Among Relatives at Risk of Lynch Syndrome
Brief Title: Initial Testing of a Behavioral Intervention About Genetic Services for Families at Risk of Lynch Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Haoyang Yan, assistant professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB-300014784; R00CA277584 (NIH)
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cascade Testing; Lynch Syndrome; Decision Making; Colorectal Cancer; Uterine Cancer; Cancer Prevention
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information Letter (Active Comparator): This arm provides an information letter about Lynch syndrome and genetic services.
  Interventions: Behavioral: Information Letter
- Information Letter and Booklet (Experimental): This arm provides an information letter with a booklet about Lynch syndrome and genetic services.
  Interventions: Behavioral: Information Letter and Booklet

INTERVENTIONS:
Behavioral: Information Letter and Booklet — an information letter with a booklet for at-risk families highlighting implications of family history, testing considerations, steps for genetic testing, and potential costs.
  Arms: Information Letter and Booklet
Behavioral: Information Letter — an information letter with basic information about LS and implications of counseling and testing of LS, and a few websites for more information and locating genetic counselors.
  Arms: Information Letter

SUMMARY:
The purpose of the study is to see if our education materials help people at risk for Lynch syndrome decide about seeking genetic services. Untested relatives of patients with Lynch syndrome will be recruited to complete a baseline survey and will be randomized to receive either the an information letter or an information letter plus a booklet. Two follow-up surveys will be administered over the span of 6 months. Participants will also be invited to join an optional exit interview to provide feedback.

DETAILED DESCRIPTION:
Lynch syndrome runs in families. It increases the risk of many types of cancer. Pre-test genetic counseling is an opportunity for at-risk people to determine whether genetic testing is right for them. Genetic testing looks for harmful changes in the genes known to cause Lynch syndrome. However, Lynch syndrome is underdiagnosed and uptake of genetic counseling and testing is low, missing opportunities for cancer prevention and early treatment.

This study is a 2-arm randomized controlled pilot trial. We aim to recruit 48 relatives at risk of LS (from about 137 probands) and randomize them to receive either the an information letter or an information letter plus a booklet. Only one relative will be enrolled per family. The primary aim of this pilot trial is to evaluate and optimize feasibility of the trial methods and the education materials to prepare for a fully powered randomized controlled trial. A brief exit interview will be conducted at 6-months post-randomization to gather any feedback about the study methods. Reasons of those who refuse to participate or drop out of the study will be assessed throughout the study.

ELIGIBILITY:
Probands Inclusion Criteria:

* English speaking
* at least 18 years old
* have had genetic testing for Lynch syndrome (LS)
* do not have a condition that would interfere with their ability to provide informed consent and complete study activities (e.g., cognitive dysfunction evaluated using clinical judgment during screening)

Clinical Trial Participants Inclusion Criteria:

* English-speaking
* at least 18 years old
* a blood relative of a patient who was diagnosed with LS
* potentially at risk for LS
* have not scheduled or had pre-test genetic counseling or genetic testing for LS
* do not have a personal history of a cancer (excluding non-melanoma skin cancer)
* do not have a condition that would interfere with their ability to provide informed consent and complete study activities (e.g., cognitive dysfunction evaluated using clinical judgment during screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment and retention rates, completeness of assessment data) | (recruitment) baseline, 1-month and 6-months post-randomization
  Record the numbers of probands approached, probands enrolled, probands who provide contact information of at least one potentially eligible relative, relatives approached, enrolled, and completing each phase of the study.
  Calculate the percentage of complete data for those participants who complete each assessment period.
Use and attitudes towards the education materials | 1-month post-randomization (may also include in 6-month post-randomization
  Assess the extent to which participants reviewed the information letter and booklet and their attitudes, likelihood of sharing the materials, feedback on the materials and impact on decisions, how the information should be delivered.
Scheduling and attendance of pre-test genetic counseling and/or genetic testing | 6-months post-randomization
  Record whether participants scheduled or attended pre-test genetic counseling and genetic testing to calculate the proportion of genetic services uptake.

SECONDARY OUTCOMES:
Scheduling and attendance of pre-test genetic counseling and/or genetic testing | 1-month post-randomization
  Record whether participants scheduled or attended pre-test genetic counseling and genetic testing to calculate the proportion of genetic services uptake.

OTHER OUTCOMES:
Psychosocial outcomes | baseline, 1-month post-randomization, 6-month post-randomization
  perceived risk, stress, fear, and coping of LS, cancer worry, colonoscopy experience, family communication, decision conflict, factors influencing decisions, self-efficacy, information received, experience and perception of facilitators and barriers of seeking genetic services for LS, perceived stress, knowledge about LS and genetic services

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No